CLINICAL TRIAL: NCT05951153
Title: Phase I, Single-arm, Dose-escalation Trial of Tributyrin to Promote Gut Health Among Children Undergoing Hematopoietic Cell Transplantation
Brief Title: Tributyrin to Promote Gut Health Among Children Undergoing Hematopoietic Cell Transplantation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI withdrew study
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00112603
Record Dates: First submitted 2023-06-26; First posted 2023-07-18 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hematopoietic Cell Transplantation (HCT)
MeSH Terms: interventions — tributyrin; Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tributyrin nutritional supplement (Experimental): Children between the ages of 2-17 with planned allogeneic hematopoietic cell transplantation with myeloablative preparative regimen, who also have standard of care nasogastric tube placement or existing gastric tubes will receive a daily dose of tributyrin.
  Interventions: Combination Product: Tributyrin

INTERVENTIONS:
Combination Product: Tributyrin — Tributyrin is a nutritional supplement prepared by esterification of glycerin with butyric acid that promotes delivery of free butyrate to distal portions of the gut.
  Other Names: Nutritional supplement

SUMMARY:
To determine the safety and tolerability of tributyrin among children undergoing hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
Primary Objectives:

1. Evaluate the safety and tolerability of tributyrin and determine the maximum tolerated dose MTD among children undergoing hematopoietic cell transplantation (HCT).

Secondary Objectives:

1. Determine the effect of tributyrin administration on fecal butyrate concentrations.
2. Measure the effect of tributyrin on gut microbiome composition and measures of gut inflammation and barrier integrity.

Hypotheses

1. Enteral administration of tributyrin will be safe and well-tolerated in children undergoing HCT at doses up to 100 mg/kg/day, with no identified dose-limiting toxicities. The most common adverse events will be gastrointestinal and will occur at frequencies and grades typically observed among children after HCT. No adverse effects will occur that are classified as probably or definitely related to the study product.
2. Tributyrin will result in a dose-dependent increase in fecal butyrate concentrations, with maximal fecal butyrate concentrations exceeding concentrations in baseline fecal samples by at least two-fold in >50% of subjects at all evaluated tributyrin doses.
3. Compared to historical controls, children receiving tributyrin will have greater preservation of gut microbial diversity and higher abundances of Clostridiales and other putatively beneficial gut anaerobes (e.g., Bifidobacterium, Lactobacillus) after HCT. Additionally, children receiving tributyrin will have lower fecal levels of calprotectin and lactoferrin and lower plasma levels of lipopolysaccharide-binding protein and intestinal fatty acid-binding protein, corresponding to lower levels of intestinal inflammation and improved gut barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-17 years with standard of care nasogastric tube placement or existing gastric tubes
* Planned allogeneic hematopoietic cell transplantation with myeloablative preparative regimen
* Planned graft-versus-host-disease prophylaxis with calcineurin inhibitor + mycophenoalte mofetil or calcineurin inhibitor + methotrexate

Exclusion Criteria:

* Previous history of hematopoietic cell transplantataion

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of tributyrin among children undergoing hematopoietic cell transplantation (HCT) | 36 months
  An evaluation of the safety and tolerability of tributyrin.

SECONDARY OUTCOMES:
Change in fecal butyrate concentration | Baseline, 36 months
Change in gut microbiome composition | Baseline, 36 months
Change in gut inflammation | Baseline, 36 months
Change in gut barrier integrity | Baseline, 36 months

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan is undecided by study team at this time.